CLINICAL TRIAL: NCT00636272
Title: Longitudinal Surveillance Registry
Acronym: LSR
Status: Terminated | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Boston Scientific CRM, Boston Scientific CRM
Other Study IDs: CR-CA-011608-T
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2008-08

CONDITIONS: Heart Failure; Sudden Cardiac Death
Keywords: ICD; CRT-D
MeSH Terms: conditions — Heart Failure; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Boston Scientific CRM's Longitudinal Surveillance Registry (LSR) will serve as an active ongoing source of updated information on the long-term reliability and performance of BSC commercially available leads and LATITUDE-enabled (wireless or wanded) pulse generators (PGs).

DETAILED DESCRIPTION:
The LSR is an active, prospective, non-randomized, multi-center registry of patients implanted with BSC commercially available LATITUDE-enabled products. The primary purpose of the LSR is to evaluate and report on the long-term reliability and clinical performance of BSC's commercially available PGs and leads using the LATITUDE Patient Management system to augment information collected from in-clinic visits. The LSR is designed to enroll patients implanted with BSC LATITUDE-enabled (wireless or wanded) commercially available PGs (lead systems may include other manufacturers' leads).

The primary objective of the LSR is to prospectively evaluate market-released PGs and leads to verify long-term system performance. The secondary objectives of the LSR include:

I. To compare PG- and lead-related reliability data collected via LATITUDE with PG- and lead-related reliability data collected at in-clinic visits II. To compare this active surveillance of BSC PG and lead reliability data to the current passive surveillance system III. To enhance understanding of feature performance, patient management and clinical outcomes

ELIGIBILITY:
Inclusion Criteria:

* Patient who is or is scheduled to be implanted within 30 days of signing the consent with a currently available BSC PG (lead systems may include other manufacturers' leads) that can be followed on the LATITUDE Patient Management system
* Patient who plans to remain in the long-term care of his/her enrolling physician (must be followed in-clinic at least once every 24 months by his/her enrolling physician)
* Patient who confirms that s/he has a telephone line compatible with the LATITUDE Patient Management system Communicator
* Patient or appropriate legal representative who is willing and capable of providing authorization for participation in the LSR

Exclusion Criteria:

* Patient who cannot be followed on the LATITUDE Patient Management system
* Patient who is unable or unwilling to comply with the protocol requirements

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient who are or will be implanted with a LATITUDE-enabled pulse generator (ICD or CRT-D).
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2008-03

CONTACTS AND LOCATIONS:
Overall Officials: Boston Scientific, Study Director — Boston Scientific Corporation